CLINICAL TRIAL: NCT06779344
Title: Myxovirus Resistance Protein a and C-Reactive Protein-Guided Antimicrobial Treatment in Outpatients with Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: MxA and CRP-Guided Use of Antimicrobial Agents for AECOPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAP-China AECOPD-bundle
Record Dates: First submitted 2024-12-23; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Acute Exacerbation Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MxA and CRP-guided group (Experimental): Perform MxA and CRP test; Report MxA and CRP results to attending clinicians; Provide MxA and CRP-based guidelines for antimicrobial treatment to the attending clinicians; Conduct follow-up telephone visits on Day 14, Day 30, and Day 90
  Interventions: Other: MxA and CRP tests; Other: MxA and CRP feedback; Other: Follow up
- Usual-care group (Active Comparator): Conduct follow-up telephone visits on Day 14, Day 30, and Day 90.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: MxA and CRP tests — A whole blood sample will be collected on the day of randomization for MxA and CRP testing.
  Arms: MxA and CRP-guided group
Other: MxA and CRP feedback — MxA and CRP results will be reported to the attending physcian within 4 hours, along with antimicrobial treatment guidelines based on these results.
  Arms: MxA and CRP-guided group
Other: Follow up — Telephone visit will be conducted on Day 14, Day 30, and Day 90 after randomization.
  Day 14 and Day 30 follow-up: antimicrobial usage; additional medical visits, hospitalization, death, symptom scores (CAT score and mMRC score).
  Day 90 follow-up: Occurrence of another exacerbation of COPD, symptom scores (CAT score and mMRC score), death.

SUMMARY:
This randomized controlled trial will investigate the clinical impact of Myxovirus Resistance A (MxA) and C-Reactive Protein (CRP)-guided antimicrobial treatment compared to usual care in outpatients with acute exacerbations of chronic obstructive pulmonary disease (AECOPD).

DETAILED DESCRIPTION:
Respiratory viral infections are a leading cause of acute exacerbations of chronic obstructive pulmonary disease (AECOPD). However, there is currently a lack of rapid diagnostic methods to differentiate the cause of AECOPD, resulting in insufficient attention to viral-induced exacerbations, with antibiotic treatment remaining the primary treatment.

Myxovirus resistance protein A (MxA) has been identified as a potential biomarker to distinguish respiratory viral infections, while C-reactive protein (CRP) has been confirmed as a useful guide for antibiotic therapy in AECOPD.

This randomized controlled trial aims to investigate the clinical value of MxA and CRP-guided antimicrobial treatment in outpatients with AECOPD, with the goal of reducing antibiotic overuse and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years old；
* Current or former smoker with a minimum smoking history of 10 pack years, clinical diagnosed with mild-to-severe COPD;
* Presenting with an acute exacerbation of COPD
* The severity of AECOPD is mild to moderate.

Exclusion Criteria:

* Required urgent hospitalization
* Received interferon therapy within 30 days before screening
* Had an active systemic inflammatory condition within 30 days prior to screening, such as cerebral infarction, myocardial infarction, or surgery
* Received vaccine in the past 30 days
* Active tuberculosis
* Immunocompromised
* Presenting with current respiratory failure
* Clinical suspicion of pneumonia or pulmonary edema.
* Coexisting bronchiectasis, cystic fibrosis, or asthma
* Had a concurrent infection at another site, such as urinary tract infections or sinusitis;
* Contraindications to antibiotics and/or antivirals
* Known etiology of the present exacerbation
* Pre-treatment with corticosteroids (cumulative dose of methylprednisolone ≥ 80 mg or equivalent dose) for the present exacerbation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day treatment failure rate | 30 days
  Defined as the proportion of patients who had additional medical visits, hospitalization, or death by Day 30.

SECONDARY OUTCOMES:
30-day hospitalization rate | 30 days
  Defined as the proportion of patients who were hospitalized by day 30
14-day treatment failure rate | 14 days
  Defined as the proportion of patients who had additional medical visits, hospitalization, or death by Day 14.
The rate of antibiotic prescriptions | 24 hours
  Defined as the proportion of patients who were prescribed antibiotics within 24 hours after randomization
The rate of antiviral prescriptions | 24 hours
  Defined as the proportion of patients who were prescribed antiviral drugs within 24 hours after randomization.
The rate of corticosteroids prescriptions | 24 hours
  Defined as the proportion of patients who were prescribed corticosteroids within 24 hours after randomization.
30-day antibiotic use rate | 30 days
  Defined as the proportion of patients who received antibiotic treatment by Day 30.
30-day antiviral use rate | 30 days
  Defined as the proportion of patients who received antiviral treatment by Day 30
30-day corticosteroids use rate | 30 days
  Defined as the proportion of patients who received corticosteroids treatment by Day 30.
the rate of next exacerbation | 90 days
  Defined as the proportion of patients who experienced another exacerbation of COPD by day 90.

OTHER OUTCOMES:
The CAT symptom score | 14 days, 30 days, 90 days
  The COPD Assessment Test (CAT) symptom score will be measured on Days 1, 14, 30, and 90.
  CAT is used to assess the severity of symptoms in patients with COPD, ranging from 0-40, with higher scores indicating more severe symptoms.
mMRC symptom score | 14 days, 30 days, 90 days
  The modified medical research council (mMRC) will be performed on Day 1, Day 14, Day 30, and Day 90. The mMRC score is used to assess the severity of dyspnea, ranging from 0 (mildest) to 4 (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared.
Supporting Information: CSR